CLINICAL TRIAL: NCT03542097
Title: Assessment of MGMT Promoter Methylation and Clinical Benefit From Temozolomide-based Therapy in Ewing Sarcoma Patients
Brief Title: Assessment of MGMT Promoter Methylation in Advanced Ewing Sarcoma Treated With Temozolomide and Irinotecan
Acronym: MGMTLiberati
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Sponsor
Other Study IDs: TEMIRI-EW
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Ewing Sarcoma Family of Tumors
Keywords: Ewing Sarcoma
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh and Formaline Fixed Paraffin Embeded tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temozolomide and Irinotecan treatment: The group include all the patients with histological confirmed diagnosis of Ewing's Sarcoma who received chemotherapic treatment with temozolomide and irinotecan. In this group the MGMT methylation evaluation will be done
  Interventions: Other: MGMT methylation evaluation

INTERVENTIONS:
Other: MGMT methylation evaluation — The MGMT methylation will be evaluated by extracting DNA from fresh and Formalin Fixed paraffin Embedded (FFPE) tumor samples

SUMMARY:
This is a biological study in patients with advanced Ewing Sarcoma who received, according, clinical practice, temozolomide and irinotecan The O6-methylguanine-DNA methyltransferase (MGMT) methylation status, will be correlated with the disease clinical data and with the disease response

DETAILED DESCRIPTION:
This is a biological study in patients with advanced Ewing Sarcoma who received, according, clinical practice, temozolomide and irinotecan.

The MGMT methylation status will be correlated with the disease clinical data and with the disease response also in term of metabolic activity (if data will be available) The MGMT methylation analysis will be performed extracting from fresh tumor sample, the DNA on the basis of the standard protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed diagnosis of Ewing Sarcoma
2. Chemotherapic treatment with temozolomide and irinotecan
3. Written informed consent prior to any study related activities

Exclusion Criteria:

1. Lack of written informed consent for the study
2. Any situation that could interfere with the complete data collection of the clinical data related to the temozolomide and irinotecan treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with advanced Ewing Sarcoma treated in clinic
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of MGMT promoter methylation | at day 1
  Amplification the methylation-specific Polymerase Chain Reaction products will be electrophoresed on a 2% agarose gel and will visualized with UV light

SECONDARY OUTCOMES:
Correlation of the MGMT promoter methylation to the activity of the temozolomide irinotecan combination | at month 2, 4, 6, 8, 10 and 12
  Correlation with level of MGMT methylation with tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Palmerini, MD, Principal Investigator — Rizzoli Orthopedic Institute
Locations (5):
- Italy (4):
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan, Mi
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, Turin
  - Orthopedic Rizzoli Institute, Bologna
  - Ospedale infantile Regina Margherita, Turin
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No Plan

REFERENCES:
- [Background] Kushner BH, Meyers PA. How effective is dose-intensive/myeloablative therapy against Ewing's sarcoma/primitive neuroectodermal tumor metastatic to bone or bone marrow? The Memorial Sloan-Kettering experience and a literature review. J Clin Oncol. 2001 Feb 1;19(3):870-80. doi: 10.1200/JCO.2001.19.3.870. PMID 11157041
- [Background] Bacci G, Ferrari S, Longhi A, Donati D, De Paolis M, Forni C, Versari M, Setola E, Briccoli A, Barbieri E. Therapy and survival after recurrence of Ewing's tumors: the Rizzoli experience in 195 patients treated with adjuvant and neoadjuvant chemotherapy from 1979 to 1997. Ann Oncol. 2003 Nov;14(11):1654-9. doi: 10.1093/annonc/mdg457. PMID 14581274
- [Background] Casey DA, Wexler LH, Merchant MS, Chou AJ, Merola PR, Price AP, Meyers PA. Irinotecan and temozolomide for Ewing sarcoma: the Memorial Sloan-Kettering experience. Pediatr Blood Cancer. 2009 Dec;53(6):1029-34. doi: 10.1002/pbc.22206. PMID 19637327
- [Background] Donson AM, Addo-Yobo SO, Handler MH, Gore L, Foreman NK. MGMT promoter methylation correlates with survival benefit and sensitivity to temozolomide in pediatric glioblastoma. Pediatr Blood Cancer. 2007 Apr;48(4):403-7. doi: 10.1002/pbc.20803. PMID 16609952
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010

DOCUMENTS (1):
  • Study Protocol (2014-01-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT03542097/Prot_000.pdf